CLINICAL TRIAL: NCT03222713
Title: School-based Program of Promotion of Self-regulation for Healthy Eating and Oral Health: Study in the Context of the School Health Program in Brazil
Brief Title: School-based Program Promotion of Self-regulation in Eating Healthy and Oral Health
Acronym: SRH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cleidilene Ramos Magalhães, Professor, Project Coordinator Cleidilene Ramos Magalhães, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Self-regulation in health
Record Dates: First submitted 2017-05-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Self-regulation in Health
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: The participants were randomly assigned into three groups: Condition I followed the health school program (PSE), Condition II group followed the PSE and the Self-regulation Health - SRH program, and the control group did not enroll in either of the health promotion programs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Program Self-regulation in health — The intervention program with children will be run by teachers and health professionals (Condition Group II) in 50-minute biweekly sessions which will take place in class in school year. During these sessions, the children will complete the following tasks: the reading of the chapters of Yellow Trials and Tribulations (one chapter per week) and the discussions and activities related to the topics of healthy eating and oral health.

SUMMARY:
The Health and Education Ministries of Brazil launched the Health in School Program - PSE - in 2007. The purpose of the PSE is twofold: articulate the actions of the education and health systems to identify risk factors and prevent them; and promote the education for health in the public elementary school system. In the health field, the self-regulation (SR) construct can contribute to the understanding of life habits which can affect the improvement of individuals' health. This study aims to present a school-based program, Promotion of Self-Regulation in Health (SRH), which adds the self-regulation approach to the topics of healthy eating and oral health of the PSE for elementary school. A study of a randomized clinical trial enrolling the 5th grade students of public elementary schools from the south of Brazil is presented. The study has two phases. In Phase 1, teachers and health professionals will participate in a training program on SRH, and in Phase 2, they will conduct an intervention in class: Promotion of SRH. The participants were randomly assigned into three groups: Condition I followed the PSE program, Condition II group followed the PSE and the SRH program, and the control group did not enroll in either of the health promotion programs. For the evaluation of the study, the following measures and instruments were applied: Body Mass Index (BMI), Simplified Oral Hygiene Index (OHI-S), Previous Day Food Questionnaire (PFDQ), Declarative Knowledge for Health Instrument, Food Preference Instrument, Student´s Attitudes and Perceptions and Parents Perceptions and Influences on the Health Instrument, Food Availability and Oral Health Instrument, Self-Regulation for Health Scale, Self-Efficacy for Health Scale. Students in the three groups will be assessed five times throughout the year: before the beginning of the intervention program, three months into intervention, six months into intervention, at the end of the intervention, and, finally, six months post intervention to check for the impact of the program on children health.

ELIGIBILITY:
Inclusion Criteria:

* Teachers must teach a 5th grade class in a public elementary school
* Health professionals must be working in a primary care unit;
* Students must be enrolled in the 5th grade in a public elementary school;
* Parents/guardians: must be responsible for a child enrolled in a 5th grade class in a public elementary school
* All participants must be volunteers and must sign the Free and Informed Consent Term or Term of Assent (parents / guardians and students);

Exclusion Criteria:

Potential participants who do not meet all the inclusion criteria, including 5th grade students with special educational needs that limit their cognitive autonomy, will be excluded from the study

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 429 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Self-regulation skills for healthy eating and oral health | 3 years
  Development of self-regulatory competencies for healthier eating and oral health in childhood. These variables wiil be evaluated through Self-Regulation for Health Scale.
Self-efficacy perception for healthy eating and oral health | 3 years
  Develop increased self-efficacy perception for healthy eating and oral health care. These variables wiil be evaluated through Self-efficacy for Health Scale.
Declarative Knowledge for Health | 3 years
  Questions for evaluate children knowledge have about healthy eating and oral health. Will be evaluated the numbers of correct answer. These variable These variable wiil be evaluated through Declarative Knowledge for Health Instrument.

SECONDARY OUTCOMES:
Body Mass Index | 3 years
  Numbers of students with Index of overweight, obesity and thinness in the study population. These measure will be evaluated trough BMI.
Simplified Oral Hygiene Index - OHI-S | 3 years
  Numbers and classification of Index of oral hygiene (good, regular and poor), Identified by the presence of dental plaque in the study population.
Food consumption information | 3 years
  Seeks information from schoolchildren about the food they consumed on the day prior. will be evaluated the food group consumed in each meals on three days of week. These variable will evaluated by Previous Day Food Questionnaire .

CONTACTS AND LOCATIONS:
Locations (1):
- Cleidilene Ramos Magalhaes, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No